CLINICAL TRIAL: NCT02811575
Title: Type 2 Diabetes and Alteration of Immune System of Intestinal Mucosa : Proof of Concept
Acronym: SIMMUNIDIA
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/16/8217
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes
Keywords: Coloscopy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ileon and colon biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with diabetes: Patients with type 2 diabetes will have biopsy during coloscopy.
  Interventions: Other: Biopsy
- Control: Patients without type 2 diabetes will have biopsy during coloscopy.
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Ileon and colon biopsy

SUMMARY:
Type 2 diabetes is the predominant type of diabetes. Because a quiet evolution, it is difficult to have a rapid diagnose. A better knowledge about pathophysiological mechanisms at the origin of type 2 diabetes and about its complications could make it possible to improve the prevention and the treatment of this disease.

Research team developped a new research axis : the microbiota of the intestinal mucosa. They proved a translocation process of intestinal bacteria from the intestinal mucosa to different tissue of the organism implicated in glucose homeostasis. This mechanism is involved in the type 2 diabetes development. A clinical study (MICIMAB) of predictive biomarkers of diabetes and obesity is ongoing.

In parallel, the same team explored the role of intestinal immunity modifications in the bacteria translocation from the gut to the blood circulation. They already have some results on animal model but not yet in human. In animal model, a solid reduction of lymphocytes T CD4 Th17 in the intestinal wall is responsable of the translocation of intestinal bacteria and in the induction of a metabolic inflammation wich promotes insulin resistance, abdominal obesity development and type 2 diabetes.

The aim of this study is to explore this hypothesis in human to have therapeutic solution later.

ELIGIBILITY:
Inclusion Criteria:

* Coloscopy indication
* Capacity to give a written informed consent

Exclusion Criteria:

* Type 1 diabetes
* Severe renal failure
* Antecedent of liver fibrosis and/or liver failure
* Antecedent of inflammatory bowel disease, lymphocyte colitis, celiac disease or colon cancer
* Antecedent of obesity surgery or of total colectomy
* Antecedent of documented intestinal ischaemia
* Acute infection the week before the inclusion
* Congenital of acquired immune deficiency
* Chronic viral infection
* Antibiotic of probiotic the month before the coloscopy
* Pregnancy
* Patients participating to another research with an exclusion period
* Patients under guardianship

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnoses of type 2 diabetes and patient who do not have a know diabetes diagnose.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Number of lymphocyte TCD4 Th17 in colon sample | Day 1
  After colon biopsy, lymphocytes TCD4 Th17 are counted in biopsy sample.

SECONDARY OUTCOMES:
Number of lymphocyte TCD4 Th17 in ileon sample | Day 1
  After ileon biopsy, lymphocytes TCD4 Th17 are counted in biopsy sample.
Number of CD45+ cells in colon sample | Day 1
  After colon biopsy, CD45+ cells are counted in biopsy sample.
Number of CD45+ cells in ileon sample | Day 1
  After ileon biopsy, CD45+ cells are counted in biopsy sample.
Activation of CD45+ cells in colon sample | Day 1
  After colon biopsy, CD45+ cells are analysed to see their state of activation in biopsy sample.
Activation of CD45+ cells in ileon sample | Day 1
  After ileon biopsy, CD45+ cells are analysed to see their state of activation in biopsy sample.
Microbiota sequencing in blood sample | Day 1
  Microbiota will be sequencing in blood sample
Microbiota quantification in blood sample | Day 1
  Microbiota will be quantified in blood sample
Microbiota sequencing in ileon sample | Day 1
  Microbiota will be sequencing in ileon sample
Microbiota sequencing in colon sample | Day 1
  Microbiota will be sequencing in colon sample
Microbiota quantification in ileon sample | Day 1
  Microbiota will be quantified in ileon sample
Microbiota quantification in colon sample | Day 1
  Microbiota will be quantified in colon sample
Bacteria production | Day 1
  Culture of biological samples to study the bacteria production

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Gourdy, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No